CLINICAL TRIAL: NCT04260451
Title: Comparison of Postoperative Pulmonary Complications Between Driving Pressure Guided Ventilation and Conventional Protective Ventilation in Thoracic Surgery
Brief Title: Driving Pressure and Postoperative Pulmonary Complications in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Severance Hospital (Other); Seoul National University Hospital (Other); Asan Medical Center (Other); Korea University Guro Hospital (Other); The Catholic University of Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SMC2019-07-182-009
Record Dates: First submitted 2020-01-31; First posted 2020-02-07 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: One-Lung Ventilation; Postoperative Complications; Driving Pressure; Postoperative Pulmonary Complication; Thoracic Surgery; Positive End Expiratory Pressure
Keywords: Postoperative pulmonary complication; Driving pressure; Thoracic surgery; One lung ventilation; Positive end expiratory pressure
MeSH Terms: conditions — Postoperative Complications | interventions — Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Driving pressure group (Experimental): Positive end expiratory pressure is adjusted to tidal volume of 5 mL/kg of ideal body weight, inspiratory:expiratory=1:2, and minimize driving pressure (plateau pressure minus end expiratory pressure) during one-lung ventilation. Other procedures are same with the control arm.
  Interventions: Other: ventilation
- Protective Ventilation (No Intervention): The control arm receives existing conventional protective ventilation with tidal volume of 5mL/kg of ideal body weight and positive end expiratory pressure of 5cmH2O during one-lung ventilation

INTERVENTIONS:
Other: ventilation — Driving Pressure Limited Ventilation
  Positive end expiratory pressure is adjusted to minimize driving pressure, plateau pressure minus end expiratory pressure from 10 to 2 cmH2O during one-lung ventilation.
  1. Lung recruitment: stepwise increase of positive end expiratory pressure 5,10,15 cmH2O with tidal volume 5mL/kg, inspiratory:expiratory 1:1, respiratory rate 10. and driving pressure up to 20 cmH2O. Then decremental PEEP titration is performed using a volume-controlled ventilation until the lowest driving pressure (plateau pressure minus PEEP) is found. This individualized PEEP is adjusted during one-lung ventilation.
  Arms: Driving pressure group

SUMMARY:
Pulmonary complications are the most common complication in thoracic surgery and the leading cause of mortality.Therefore, lung protection is utmost important, and protective ventilation is strongly recommended in thoracic surgery. Protective ventilation is a prevailing ventilatory strategy in these days and is comprised of small tidal volume, limited inspiratory pressure, and application of positive end-expiratory pressure. However, several retrospective studies recently suggested that tidal volume, inspiratory pressure, and positive end-expiratory pressure are not related to patient outcomes, or only related when they influenced the driving pressure. Recently, the investigators reported the first prospective study about the driving pressure-guided ventilation in thoracic surgery. PEEP was titrated to bring the lowest driving pressure in each patient and applied throughout the one lung ventilation. The application of individualized PEEP reduced the incidence of pulmonary complications.However, that study was small size single center study with 312 patients. Thus, investigators try to perform large scale multicenter study. Through this study investigators evaluate that driving pressure-guided ventilation can reduce the incidence of postoperative pulmonary complications compared with conventional protective ventilation in thoracic surgery.

DETAILED DESCRIPTION:
Nowdays, the usual setting of protective ventilation during one lung ventilation is tidal volume (VT) 5 ml/kg of predicted body weight, positive end-expiratory pressure (PEEP) 5 cm H2O and plateau pressure (Pplat) less than 25 cmH2O.

However, a high incidence of postoperative pulmonary complications is still being observed even with a protective ventilatory strategy.

Driving pressure is [Pplat - PEEP] and is the pressure required for the alveolar opening. Static lung compliance (Cstat) is expressed as [VT / (Pplat - PEEP)]. Thus, driving pressure is also expressed as [VT / Cstat]. Driving pressure has an inverse relationship with Cstat and orthodromic relationship with VT according to this formula. High driving pressure indicates poor lung condition with decreased lung compliance.

Thus, investigator try to prove that driving pressure limited ventilation is superior in preventing postoperative pulmonary complications to existing protective ventilation in large scale multicenter study.

Recruit maneuver perform all group after intubation (stepwise increase of positive end expiratory pressure 5,10,15 cmH2O with tidal volume 5mL/kg).

The control arm receives existing conventional protective ventilation with tidal volume of 5mL/kg of ideal body weight and PEEP of 5 cmH2O during one-lung ventilation.

The driving pressure arm receives driving pressure limited ventilation with tidal volume of 5mL/kg of ideal body weight and individualized PEEP. Individualized PEEP is adjusted to minimize driving pressure, it find through decremental PEEP titration from 10 to 2 cmH2O during one-lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

Adults older than or equal to 19 years with American Society of Anesthesiologists physical status Ⅰ-Ⅲ Patient who undergoes one-lung ventilation (more than 60 minutes) for elective thoracic surgery

Exclusion Criteria:

1. The American Society of Anesthesiologists (ASA) Physical Status classification greater than or equal to 4
2. Symptoms of heart failure (hypertension, urination, pulmonary edema, left ventricular outflow rate <45%) or preoperative vasopressors
3. Patient who is received oxygen therapy and ventilation care
4. large emphysema and pneumothorax
5. pregnancy and lactation
6. patients participating in similar studies
7. Joint with other operation
8. Patient who rejects being enrolled in the study
9. Patients with elevated intracranial pressure
10. Patients with peripheral neuropathy or blood circulation disorders
11. Patients with hematology disease
12. Congenital heart disease with shunt

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative pulmonary complications | within the first 7 days after surgery
  Postoperative pulmonary complications are defined as one or more of the following:
  * Hypoxia: SpO2 < 90%
  * Requiring oxygen therapy: Facial mask, nasal prong, continuous positive airway pressure, non-invasive positive pressure breathing or high flow nasal oxygen supply between POD 2 and 7.
  * Initial ventilator supports longer than 24 h
  * Re-intubation
  * Requiring mechanical ventilation
  * Tracheostomy
  * Pneumonia
  * Empyema
  * Atelectasis requiring bronchoscopy
  * Acute respiratory distress syndrome
  * Acute lung injury
  * Persistent emphysema or pneumothorax or air leak requiring chest tube for 5 days or more
  * Prolonged pleural effusion requiring chest tube for 5 days or more
  * Bronchopleural fistula
  * Contralateral pneumothorax
  * Pulmonary embolism embolism

SECONDARY OUTCOMES:
oxygenation | 15 minutes after one-lung ventilation
  Partial pressure of oxygen in arterial blood (PaO2, mmHg) or PaO2/Inspired oxygen fraction (PF ratio)
the incidence of rescue ventilation | during surgery
  the need for rescue ventilation to treat hypoxia (Inspired oxygen fraction 1.0, two lung ventilation, recruitment, PEEP change, Tidal volume change, continuous positive pressure ventilation, change to pressure control mode)
Cstat | 15 minutes after one-lung ventilation
  Lung compliance (mL/mmHg)
CRP | within the first 1 days after surgery
  C-reactive protein (mg/L) of laboratory exam
the incidence of postoperative transfusion | within the first 3 days after surgery
  red blood cell, fresh frozen plasma, platelet
the incidence of postoperative renal complications | within the first 7 days after surgery
  acute kidney injury(acute kidney injury network criteria): Stage I: Diuresis < 0.5 mg/kg (6 h) or increase in serum Cr > 0.3 mg/dl. Stage II: Diuresis < 0.5 mg/kg (12 h) or basal Cr x 2 mg/dL. Stage III: Diuresis < 0.3 mg/kg (24 h) or anuria (12 h) or basal Cr x 3 mg/dL, or Cr > 4 mg/dL or renal replacement therapy.
the incidence of postoperative cognitive complications | within the first 7 days after surgery
  diagnosed by Confusion Assessment method (CAM: positive or negative) or Medicines for treating delirium symptoms include antipsychotic drugs and benzodiazepines
the incidence of postoperative surgical site complications | within the first 7 days after surgery
  : The CDC defines a superficial incisional surgical site infection as one which meets the following criteria.
  1. Infection occurs within 30 days after surgery and
  2. Involves only skin and subcutaneous tissue of the incision and
  3. The patient has at least one of the following:
     1. purulent drainage from the superficial incision
     2. organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision
     3. at least one of the following symptoms or signs of infection: pain or tenderness, localised swelling, redness or heat, and superficial incision is deliberately opened by surgeon and is culture positive or not cultured. A culture negative finding does not meet this criterion.
     4. diagnosis of an incisional surgical site infection by a surgeon or attending physician.
the incidence of acute myocardial infarction | within the first 7 days after surgery
  Acute myocardial injury with clinical evidence of acute myocardial ischemia and with detection of a rise and/or fall of cardiac troponin values with at least one value above the 99th percentile upper reference limit and at least one of the following:
  1. Symptoms of myocardial ischemia
  2. New ischemic ECG changes
  3. Development of pathological Q waves
  4. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic etiology
  5. Identification of a coronary thrombus by angiography or autopsy (not for types 2 or 3 myocardial infarctions)
the incidence of coronary thrombosis | within the first 7 days after surgery
  Percutaneous coronary intervention or coronary artery surgery
the incidence of cerebral infarction | within the first 7 days after surgery
  Magnetic resonance imaging diagnosis
the incidence of septic shock | within the first 7 days after surgery
  : A subset of sepsis (a life-threatening organ dysfunction resulting from dysregulated host responses to infection) in which underlying circulatory, cellular, and metabolic abnormalities are profound enough to substantially increase the risk of mortality. Despite adequate fluid resuscitation, patients have hypotension requiring vasopressors to maintain a mean arterial blood pressure above 65 mmHg and have an elevated serum lactate concentration of more than 2 mmol/L
the incidence of new arrythmia | within the first 7 days after surgery
  New arrhythmias that persist for more than 2 days
Length of stay in the intensive care unit and hospital | within the first 30 days after surgery
  the duration of hospital stay and intensive care unit stay (day)
the incidence of re-admission | within the first 30 days after surgery
  re-admission because of surgical related problems
mortality | within the first 30 days after surgery
  in hospital death or out of hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

REFERENCES:
- [Derived] Park M, Yoon S, Nam JS, Ahn HJ, Kim H, Kim HJ, Choi H, Kim HK, Blank RS, Yun SC, Lee DK, Yang M, Kim JA, Song I, Kim BR, Bahk JH, Kim J, Lee S, Choi IC, Oh YJ, Hwang W, Lim BG, Heo BY. Driving pressure-guided ventilation and postoperative pulmonary complications in thoracic surgery: a multicentre randomised clinical trial. Br J Anaesth. 2023 Jan;130(1):e106-e118. doi: 10.1016/j.bja.2022.06.037. Epub 2022 Aug 20. PMID 35995638